CLINICAL TRIAL: NCT04586751
Title: The Impact of Pecs Blocks on the Appearance of Post Mastectomy Chronic Pain Symptoms
Brief Title: The Impact of Pecs Blocks on Postmastectomy Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Breast-Nektaria
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Pain Syndrome; Pain, Postoperative; Chronic Pain; Breast Cancer; Breast Soft Tissue Neoplasm; Breast Neoplasms; Breast Cancer Female; Breast Pain; Anesthesia
MeSH Terms: conditions — Somatoform Disorders; Pain, Postoperative; Chronic Pain; Breast Neoplasms; Mastodynia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): Pecs block under real-time ultrasound guidance after anesthesia induction will be performed. In specific, using the in-plane insertion technique, after visualization of the entire needle as a bright hyperechoic line and aiming between pectoralis major and pectoralis minor at the 3rd rib level, 2 ml of normal saline 09% will be injected first, to verify the correct position of the needle. Followingly, 10 mL ropivacaine 0.5% will be injected in order to block the lateral and medial pectoral nerves. Finally, another 15 ml of ropivacaine 0.5% plus 4 mg of dexamethasone will be injected between the pectoralis minor muscle and the anterior serratus muscle,at the level of the 4th and 5th ribs, after negative aspiration, to block the intercostal and intercostobrachial nerves. Using the color Doppler the vessels will be identified, so that their puncture is avoided during the procedures.
  Interventions: Other: Pecs block
- control group (Sham Comparator): no regional block will be performed
  Interventions: Other: no Pecs block

INTERVENTIONS:
Other: Pecs block — Pecs block under real-time ultrasound guidance after anesthesia induction will be performed.
  Arms: study group
Other: no Pecs block — no regional block will be performed in this arm
  Arms: control group

SUMMARY:
The aim of the present study is to investigate the incidence of chronic pain following breast cancer surgery in Cyprus, discover its associated risk factors and explore the impact of Pecs Blocks on the appearance of post mastectomy chronic pain symptoms

DETAILED DESCRIPTION:
Breast cancer is the commonest type of malignancy in women. Chronic postoperative neuropathic pain may appear either in the early postoperative period or at a later stage, usually 3-6 months post-operatively. Chronic post-operative pain syndrome of any magnitude usually involves 19-57% of patients that have undergone any kind of surgical procedure, while 5% of them experience intense symptoms. Risk factors for developing post-mastectomy pain syndrome include younger age, increased Body mass Index (BMI), psychological profile, co-existence of other painful conditions, pre-operative radiotherapy/chemotherapy, type of surgical procedure and anaesthesia, persistent acute postoperative pain, etc. Consequently, chronic post mastectomy pain syndrome results in significant psychosomatic sequelae with variable social impacts for the female patients.

The aim of the present study will be to investigate the incidence of chronic pain following breast cancer surgery in Cyprus, discover its associated risk factors and explore the impact of Pecs Blocks on the appearance of post mastectomy chronic pain symptoms.

During the preoperative visit, the women will be informed about the study and will be instructed to the use of the pain numeric rating scale (NRS) graded from 0 to 10. Standardized anesthesia will be administered. All patients will receive 1000 mg of paracetamol and 0.07 mg/ Kg of morphine intraoperatively. In the Post-Anesthesia Care Unit (PACU), patients will receive additional morphine boluses on request, until NRS score is lesser or equal than 4. Postoperative nausea and vomiting will be treated with ondansetron 4 mg iv. After discharge from PACU, patients will receive a combination of paracetamol 1 gr/6h and im pethidine 75 mg on request, as per hospital protocol.

Numerical rating scores (NRS) at rest and movement will be measured at 6h, 12h and 24h postoperatively. Additionally, the time to first request for analgesia after surgery will be noted.

All patients will also be evaluated 3 and 6 months after surgery with the use of NRS at rest and movement and additionally, via the use of Douleur Neuropathique (DN4) questionnaire for the occurence of neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-III patients
* Breast cancer patients
* Patients who receive operative treatment

Exclusion Criteria:

* inability to consent to the study due to language barriers or cognitive dysfunction -
* skin infection at the puncture site
* contraindication to paracetamol administration
* known previous hepatic or renal impairment as assessed by the patients' history and routine biochemical markers

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
pain score 6 hours postoperatively | 6 hours after surgery
  pain score by the use of Numeric Rating Scale (NRS) 6 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 12 hours postoperatively | 12 hours after surgery
  pain score by the use of Numeric Rating Scale (NRS) 12 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 24 hours postoperatively | 24 hours after surgery
  pain score by the use of Numeric Rating Scale (NRS) 24 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"

SECONDARY OUTCOMES:
incidence of chronic pain | 3 months after surgery
  occurrence of chronic pain at the site of the operation 3 months after surgery, with the use of the Numeric Rating Scale (NRS), at rest and during movement
incidence of chronic pain | 6 months after surgery
  occurrence of chronic pain at the site of the operation 6 months after surgery, with the use of the Numeric Rating Scale (NRS), at rest and during movement
time of first request for analgesia | 24 hours postoperatively
  time of first request for analgesia after the operation
analgesic consumption in mg of morphine | 24 hours postoperatively
  additional analgesic consumption in the first 24 hours after the operation
satisfaction from postoperative analgesia | 24 hours postoperatively
  satisfaction from postoperative analgesia on a four-point Likert scale with 1 marked as minimal satisfaction and 4 as maximal satisfaction
Pecs block related complications | 48 hours postoperatively
  Pecs block-related complications at the site of the local anesthetic injection

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, Principal Investigator — Aretaieion University Hospital
Locations (3):
- Cyprus (2):
  - General Hospital of Limassol, Limassol
  - General Hospital of Nicosia, Nicosia
- Aretaieion University Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bashandy GM, Abbas DN. Pectoral nerves I and II blocks in multimodal analgesia for breast cancer surgery: a randomized clinical trial. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):68-74. doi: 10.1097/AAP.0000000000000163. PMID 25376971
- [Background] Thomas M, Philip FA, Mathew AP, Jagathnath Krishna KM. Intraoperative pectoral nerve block (Pec) for breast cancer surgery: A randomized controlled trial. J Anaesthesiol Clin Pharmacol. 2018 Jul-Sep;34(3):318-323. doi: 10.4103/joacp.JOACP_191_17. PMID 30386013
- [Background] Sykioti P, Zis P, Vadalouca A, Siafaka I, Argyra E, Bouhassira D, Stavropoulou E, Karandreas N. Validation of the Greek Version of the DN4 Diagnostic Questionnaire for Neuropathic Pain. Pain Pract. 2015 Sep;15(7):627-32. doi: 10.1111/papr.12221. Epub 2014 May 5. PMID 24796220
- [Background] Bras M, Dordevic V, Gregurek R, Bulajic M. Neurobiological and clinical relationship between psychiatric disorders and chronic pain. Psychiatr Danub. 2010 Jun;22(2):221-6. PMID 20562750
- [Background] Dujmovic A, Marcinko D, Bulic K, Kisic H, Dudukovic M, Mijatovic D. Quality of Life and Depression Among Female Patients Undergoing Surgical Treatment for Breast Cancer: A Prospective Study. Psychiatr Danub. 2017 Sep;29(3):345-350. doi: 10.24869/psyd.2017.345. PMID 28949315
- [Background] Khan RS, Ahmed K, Blakeway E, Skapinakis P, Nihoyannopoulos L, Macleod K, Sevdalis N, Ashrafian H, Platt M, Darzi A, Athanasiou T. Catastrophizing: a predictive factor for postoperative pain. Am J Surg. 2011 Jan;201(1):122-31. doi: 10.1016/j.amjsurg.2010.02.007. Epub 2010 Sep 15. PMID 20832052
- [Background] Najeeb HN, Mehdi SR, Siddiqui AM, Batool SK. Pectoral Nerves I, II and Serratus Plane Blocks in Multimodal Analgesia for Mastectomy: A Randomised Clinical Trial. J Coll Physicians Surg Pak. 2019 Oct;29(10):910-914. doi: 10.29271/jcpsp.2019.10.910. PMID 31564259
- See also: contains news, features and comments on every topic that matters to the pain community — http://www.painconcern.org.uk